CLINICAL TRIAL: NCT03527719
Title: Effectiveness of a Standardized Protocol-based Treatment Program on Hypertension Control in Rural China
Brief Title: China Rural Hypertension Control Project
Acronym: CRHC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Hospital of China Medical University (Other)
Collaborators: Tulane University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Tongji Hospital (Other); Disease Control and Prevention Centre of Liaoning Province (Unknown); Chaoyang Central Hospital (Other); Hanzhong People's Hospital (Unknown); Disease Control and Prevention Centre of Chaoyang City (Unknown); Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yingxian Sun, Chief of Department of Cardiology in First Hospital of China Medical University, First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KLS20181582
Record Dates: First submitted 2018-04-22; First posted 2018-05-17 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-08

CONDITIONS: Hypertension
Keywords: Hypertension; Cardiovascular disease; Dementia; China; Protocol-based treatment; Stroke
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Dementia; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessment Committee members will be blinded to outcome assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Village-doctor-led multifaceted intervention
  Interventions: Other: Village-doctor-led multifaceted intervention
- Control Group (No Intervention): Village doctors in usual care group will not receive hypertension management training or support. However, they will be trained in standardized BP measurement. Participants in control group will receive their usual care from village doctors or primary care physicians in township hospitals

INTERVENTIONS:
Other: Village-doctor-led multifaceted intervention — * Establishing a network including hypertension specialists at city/county hospitals, primary care physicians at township hospitals, and village doctors to collaboratively manage hypertension
  * Using hypertension control rate as one of the metrics for incentive supplements to village doctors
  * Providing discounted or free antihypertensive medications to patients with hypertension
  * Training village doctors to measure blood pressure according to a standard protocol
  * Training village doctors to use a simple stepwise protocol for hypertension treatment
  * Training village doctors to conduct health coaching on lifestyle change (e.g., lowering sodium and alcohol intake) and medication adherence
  * Providing free blood-pressure monitor and training to patients for home blood pressure measurement
  * Encouraging lifestyle change and medication adherence
  * Connecting patients through WeChat or telephone for group social support
  Arms: Experimental Group

SUMMARY:
China Rural Hypertension Control (CRHC) Project is a cluster randomized trial that will test the effectiveness of a village doctor-led multifaceted intensive blood pressure intervention on hypertension control in 18 months (Phase 1), cardiovascular disease risk in 36 months (Phase 2), and all-cause dementia in 48 months (Phase 3) among patients with hypertension in rural China. An extended observational follow-up, the CRHCP post-intervention observational follow-up study, will be conducted at Year 7 to evaluate long-term effects.

DETAILED DESCRIPTION:
The overall objective of the CRHC Project is to develop an effective, adoptable, and sustainable implementation strategy to achieve more intensive blood pressure (BP) control among rural residents in China. Moreover, this effectiveness-implementation trial will test the effectiveness of a lower BP target (<130/80 mmHg) on cardiovascular disease (CVD) and all-cause dementia. Specifically, we will test the effectiveness of a village doctor-led multifaceted intervention, compared with usual care, on BP control, CVD, and dementia among rural residents with hypertension in China. This cluster randomized trial is conducted in 326 villages from three provinces in mainland China. A total of 163 villages was randomly assigned to a village doctor-led multifaceted intervention and 163 villages to usual care, stratified by provinces, counties, and townships. A total of 33,995 individuals aged ≥40 years with uncontrolled hypertension were recruited into the study. The village doctor-led multifaceted intervention is designed to overcome barriers at the healthcare system, provider, patient, and community levels. Study participants are followed every 6 months for BP, CVD, and other study outcomes. The primary outcome is BP control (<130/80 mm Hg) at 18 months in phase 1, CVD events over 36 months in phase 2, and all-cause dementia at 48 months in phase 3. In addition, an extended observational follow-up will be conducted at Year 7 without further active intervention, to evaluate long-term outcomes including major cardiovascular events, dementia or cognitive outcomes, all-cause mortality, renal outcomes, and the sustainability of implementation fidelity.

ELIGIBILITY:
Eligibility criteria for study villages:

* The village has a regular village doctor who is willing to participate in the hypertension control project
* The village does not plan to merge with other villages within 3 years
* The village is at least 2 kilometers away from other participating villages
* The village participates in the China New Rural Cooperative Medical Scheme

Eligibility criteria of study participants:

* Men or women aged ≥40 years
* Mean untreated systolic BP ≥140 mm Hg and/or diastolic BP ≥90 mm Hg or mean treated systolic BP ≥130 mm Hg and/or diastolic BP ≥80 mm Hg for individuals without a history of clinical CVD; or mean treated/untreated systolic BP ≥130 mm Hg and/or diastolic BP ≥80 mm Hg for individuals with a history of clinical coronary heart disease, heart failure, stroke, diabetes, or chronic kidney disease
* Have lived in a participating village for at least 6 months
* No intention to migrate within next 3 years
* Taking part in the New Rural Cooperative Medical Scheme
* Not pregnant or planning to become pregnant
* No malignant tumors and life expectancy ≥3 years
* Willing to participate and able to sign informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33995 (Estimated)
Dates: Start 2018-05-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome of Phase 1: Hypertension control rate | 18 months after baseline
  The proportion of participants with controlled blood pressure（< 130/80 mm Hg）
Primary Outcome of Phase 2: Composite cardiovascular disease outcome | 36 months after baseline
  Record the occurrence of newly diagnosed composite cardiovascular disease
Primary Outcome of Phase 3: All-cause dementia | 48 months after baseline
  Record all-cause dementia
Primary Outcome of Extension Study: Composite cardiovascular disease outcome | Year 7 after baseline
  Record the occurrence of newly diagnosed composite cardiovascular disease

SECONDARY OUTCOMES:
Secondary Outcome of Phase 1: Mean systolic and diastolic pressure changes | 18 months after baseline
  Mean systolic and diastolic pressure changes of participants
Secondary Outcome of Phase 1: Hypertension control rate（<140/90 mm) | 18 months after baseline
  The proportion of participants with controlled blood pressure（< 140/90 mm Hg）
Secondary Outcome of Phase 1: Adherence to antihypertensive medication rate | 18 months after baseline
  Use questionnaires to assess the proportion of participants who adhere to antihypertensive drugs
Secondary Outcome of Phase 2: Stroke | 36 months after baseline
  Number of newly diagnosed stroke
Secondary Outcome of Phase 2: Myocardial infarction | 36 months after baseline
  Number of newly diagnosed myocardial infarction
Secondary Outcome of Phase 2: Heart failure requiring hospitalization or treatment | 36 months after baseline
  Number of patients with newly diagnosed heart failure requiring hospitalization or treatment
Secondary Outcome of Phase 2: Cardiovascular disease death | 36 months after baseline
  Number of cardiovascular disease death
Secondary Outcome of Phase 2: All-cause death | 36 months after baseline
  Number of all-cause death
Secondary Outcome of Phase 2: Mean systolic and diastolic pressure changes | 36 months after baseline
  Mean systolic and diastolic pressure changes of participants
Secondary Outcome of Phase 3: Cognitive impairment no dementia | 48 months after baseline
  Record cognitive impairment no dementia
Secondary Outcome of Phase 3: Composite outcome of dementia and cognitive impairment no dementia | 48 months after baseline
  Record the composite outcome of dementia and cognitive impairment no dementia
Secondary Outcome of Phase 3: Death from all causes | 48 months after baseline
  Record death from all causes
Secondary Outcome of Phase 3: Composite outcome of dementia or deaths | 48 months after baseline
  Record the composite outcome of dementia or deaths
Secondary Outcome of Phase 3: Composite and individual cardiovascular disease (myocardial infarction, stroke, heart failure requiring hospitalization or treatment, and cardiovascular death) | 48 months after baseline
  Record the composite and individual cardiovascular disease (myocardial infarction, stroke, heart failure requiring hospitalization or treatment, and cardiovascular death)
Secondary Outcome of Phase 3: Changes in mean systolic and diastolic blood pressure from baseline to 48 months | 48 months after baseline
  Record changes in mean systolic and diastolic blood pressure from baseline to 48 months
Secondary Outcome of Phase 3: Proportion of hypertension control (BP <130/80 mm Hg or <140/90 mmHg) at 48 months | 48 months after baseline
  Record the proportion of hypertension control (BP <130/80 mm Hg or <140/90 mmHg) at 48 months
Secondary Outcome of Extension Study: Composite outcome of dementia and cognitive impairment no dementia | Year 7 after baseline
  Record the composite outcome of dementia and cognitive impairment no dementia
Secondary Outcome of Extension Study: Stroke | Year 7 after baseline
  Number of newly diagnosed stroke
Secondary Outcome of Extension Study: Myocardial infarction | Year 7 after baseline
  Number of newly diagnosed myocardial infarction
Secondary Outcome of Extension Study: Heart failure requiring hospitalization or treatment | Year 7 after baseline
  Number of patients with newly diagnosed heart failure requiring hospitalization or treatment
Secondary Outcome of Extension Study: Cardiovascular disease death | Year 7 after baseline
  Number of cardiovascular disease death
Secondary Outcome of Extension Study: All-cause death | Year 7 after baseline
  Number of all-cause death
Secondary Outcome of Extension Study: All-cause dementia | Year 7 after baseline
  Record all-cause dementia
Secondary Outcome of Extension Study: Cognitive impairment no dementia | Year 7 after baseline
  Record cognitive impairment no dementia
Secondary Outcome of Extension Study: Mean systolic and diastolic pressure changes | Year 7 after baseline
  Record changes in mean systolic and diastolic blood pressure
Secondary Outcome of Extension Study: Proportion of hypertension control (BP <130/80 mm Hg or <140/90 mmHg) | Year 7 after baseline
  Record the proportion of hypertension control (BP <130/80 mm Hg or <140/90 mmHg)
Secondary Outcome of Extension Study: Adherence to antihypertensive medication rate | Year 7 after baseline
  Use questionnaires to assess the proportion of participants who adhere to antihypertensive drugs

CONTACTS AND LOCATIONS:
Overall Officials: Yingxian Sun, MD, PhD, Principal Investigator — First Hospital of China Medical University
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun G, Ye N, Wang C, Liu S, Miao W, Qiao L, Ouyang N, Geng D, Shi C, Zhang L, Zhang P, Yin Y, Xie Z, Yu Y, Sun Y. Evaluating intensive blood pressure control versus usual care on cardiovascular disease in patients with diabetes using win statistics: a subgroup analysis of a cluster randomized trial. J Adv Res. 2025 Sep 29:S2090-1232(25)00758-1. doi: 10.1016/j.jare.2025.09.054. Online ahead of print. PMID 41033581
- [Derived] Lu X, Wang J, Chen S, Lv L, Yu J. Effect of Comprehensive Health Management on Medication Adherence and Healthy Lifestyle Behavior of Patients With Hypertension. Int J Hypertens. 2025 Jul 19;2025:1165809. doi: 10.1155/ijhy/1165809. eCollection 2025. PMID 41018530
- [Derived] Sun G, Miao W, Liu S, Yin Y, Geng D, Ye N, Xie Z, Zhang L, Zhou S, Wang C, Qiao L, Pei S, Ouyang N, Shi C, Guo X, Sun Y. Intensive Systolic Blood Pressure Reduction and Kidney and Cardiovascular Outcomes: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Jul 1;8(7):e2519604. doi: 10.1001/jamanetworkopen.2025.19604. PMID 40643915
- [Derived] He J, Zhao C, Zhong S, Ouyang N, Sun G, Qiao L, Yang R, Zhao C, Liu H, Teng W, Liu X, Wang C, Liu S, Chen CS, Williamson JD, Sun Y. Blood pressure reduction and all-cause dementia in people with uncontrolled hypertension: an open-label, blinded-endpoint, cluster-randomized trial. Nat Med. 2025 Jun;31(6):2054-2061. doi: 10.1038/s41591-025-03616-8. Epub 2025 Apr 21. PMID 40258956
- [Derived] Sun G, Guo X, Li G, Zhang P, Yin Y, Qiao L, Ye N, Wang C, Liu S, Geng D, Miao W, Xie Z, Yu Y, Li Z, Jiang X, Tan X, Sun Y. Intensive Blood Pressure Strategy on Cardiovascular Diseases in Patients With Metabolic Syndrome: Post Hoc Analysis of a Clinical Trial. J Am Heart Assoc. 2025 Mar 18;14(6):e036820. doi: 10.1161/JAHA.124.036820. Epub 2025 Mar 13. PMID 40079319
- [Derived] Sun G, Wang C, Ye N, Shi C, Ouyang N, Qiao L, Li G, Zhang L, Yu Y, Li Z, Zhou Y, Chen Z, Zhang S, Zhang P, Geng D, Miao W, Liu S, Sun Y. Impact of baseline cardiovascular risk on the outcomes of intensive blood pressure intervention: a post hoc analysis of the China rural hypertension control project. BMC Med. 2024 Jun 20;22(1):258. doi: 10.1186/s12916-024-03494-w. PMID 38902731
- [Derived] Guo X, Ouyang N, Sun G, Zhang N, Li Z, Zhang X, Li G, Wang C, Qiao L, Zhou Y, Chen Z, Shi C, Liu S, Miao W, Geng D, Zhang P, Sun Y; CRHCP Study Group. Multifaceted Intensive Blood Pressure Control Model in Older and Younger Individuals With Hypertension: A Randomized Clinical Trial. JAMA Cardiol. 2024 Sep 1;9(9):781-790. doi: 10.1001/jamacardio.2024.1449. PMID 38888905
- [Derived] He J, Ouyang N, Guo X, Sun G, Li Z, Mu J, Wang DW, Qiao L, Xing L, Ren G, Zhao C, Yang R, Yuan Z, Wang C, Shi C, Liu S, Miao W, Li G, Chen CS, Sun Y; CRHCP Study Group. Effectiveness of a non-physician community health-care provider-led intensive blood pressure intervention versus usual care on cardiovascular disease (CRHCP): an open-label, blinded-endpoint, cluster-randomised trial. Lancet. 2023 Mar 18;401(10380):928-938. doi: 10.1016/S0140-6736(22)02603-4. Epub 2023 Mar 2. PMID 36871573
- [Derived] Sun Y, Mu J, Wang DW, Ouyang N, Xing L, Guo X, Zhao C, Ren G, Ye N, Zhou Y, Wang J, Li Z, Sun G, Yang R, Chen CS, He J; CRHCP Study Group. A village doctor-led multifaceted intervention for blood pressure control in rural China: an open, cluster randomised trial. Lancet. 2022 May 21;399(10339):1964-1975. doi: 10.1016/S0140-6736(22)00325-7. Epub 2022 Apr 29. PMID 35500594
- [Derived] Sun Y, Li Z, Guo X, Zhou Y, Ouyang N, Xing L, Sun G, Mu J, Wang D, Zhao C, Wang J, Ye N, Zheng L, Chen S, Chang Y, Yang R, He J. Rationale and Design of a Cluster Randomized Trial of a Village Doctor-Led Intervention on Hypertension Control in China. Am J Hypertens. 2021 Aug 9;34(8):831-839. doi: 10.1093/ajh/hpab038. PMID 33605981